CLINICAL TRIAL: NCT07280507
Title: Comparative Evaluation of Microneedling With Injectable PRF and Hyaluronic Acid for Papilla Reconstruction: A Randomized Clinical Trial
Brief Title: Comparing Microneedling and Injectable Platelet Rich Fibrin to Hyaluronic Acid In Papilla Reconstruction
Acronym: (PRF) (HA)
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Amal Jamjoom, BDS, MS., Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 117-10-24; 117-10-24 (Registry Identifier: 117-10-24); 117-10-24 (Other: King AbdulAziz University); King AbdulAziz University (Other: King AbdulAziz University)
Record Dates: First submitted 2025-11-26; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Papilla Reconstruction
Keywords: Papilla; Reconstruction; Hyaluronic Acid; Injectable Platelet Rich Fibrin; Microneedling
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HA (Experimental): Hyaluronic Acid Filler
  Interventions: Other: Hyaluronic Acid (HA)
- iPRF (Active Comparator)
  Interventions: Biological: Injectable Platelet Rich Fibrin

INTERVENTIONS:
Biological: Injectable Platelet Rich Fibrin — Injectable Platelet Rich Fibrin
  Arms: iPRF
Other: Hyaluronic Acid (HA) — Filler
  Arms: HA

SUMMARY:
This randomized split-mouth clinical trial aims to compare the clinical effectiveness of microneedling combined with injectable platelet-rich fibrin (i-PRF) versus hyaluronic acid (HA) gel injection in the reconstruction of Class I interdental papilla loss. The study hypothesizes that MN + i-PRF will yield greater papillary regeneration, offering a minimally invasive, biologically active alternative to traditional surgical approaches for soft-tissue esthetic rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Plaque index <1
* Gingival index <1
* Class I papillary loss (Nordland and Tarnow classification)
* Probing depth ≤4 mm at the test site
* Inter-proximal bone crest distance ≤7 mm from the contact point.

Exclusion Criteria:

* Pregnancy
* Lactation
* Uncontrolled systemic diseases (e.g., diabetes)
* Anticoagulant therapy
* Recent radiotherapy
* Orthodontic treatment
* Midline diastema
* High frenum attachment
* Class II/III papillary loss.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Papillary height | Baseline, 6 weeks, and 12 weeks.
  from the mucogingival junction to the papilla tip
Papillary width | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- King AbdulAziz University, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR
Time Frame: March 2026- March 2027.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-12-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT07280507/Prot_SAP_000.pdf